CLINICAL TRIAL: NCT03668821
Title: Vascular Frailty - An Observational Cohort Study
Brief Title: Frailty in Vascular Patients Undergoing Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 18HH4445
Record Dates: First submitted 2018-09-04; First posted 2018-09-13 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Vascular Diseases; Carotid Artery Diseases; Aneurysmal Disease; Peripheral Artery Disease
Keywords: Vascular Diseases; Peripheral Artery Disease
MeSH Terms: conditions — Vascular Diseases; Carotid Artery Diseases; Peripheral Arterial Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Carotid Artery Disease: Patients with Carotid Artery Disease. Quality of life and frailty questionnaires
  Interventions: Other: Questionnaire
- Aneurysmal Disease: Patients with Aneurysmal Disease. Quality of life and frailty questionnaires
  Interventions: Other: Questionnaire
- Peripheral Artery Disease: Patients with Peripheral Artery Disease. Quality of life and frailty questionnaires
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Quality of life and frailty questionnaires

SUMMARY:
An observational cohort study of the frailty of vascular surgery patients undergoing intervention and their outcomes.

DETAILED DESCRIPTION:
Vascular surgical operations are major procedures with significant associated morbidity and mortality. Frailty is a major factor influencing surgical outcome, but the effect on morbidity/mortality and quality of life is poorly understood in vascular surgery. Activity levels play a significant role in frailty and in pre-intervention preparation. It is anticipated that as frailty levels increase, activity levels decrease. It is hypothesised that vascular surgery patients suffer from a high prevalence of frailty and that increasing frailty will lead to increased morbidity and mortality and decreased quality of life.

This initial study will provide the foundations to identify targets for improvement in degree of frailty, appropriateness for surgery and outcome.

This project aims to:

Assess and quantify the prevalence of frailty as well as recording activity levels in the vascular surgery patient cohort Explore the impact of frailty and pre-op activity on surgical outcomes in the vascular surgical patient cohort to guide surgical treatments as well as future studies aimed at improving frailty and activity and thereby quality of life.

Identification of an appropriate metric of frailty for this population group to include activity, is a secondary aim of this proposal.

ELIGIBILITY:
Inclusion Criteria:

1. All patients attending for aortic aneurysm repair, carotid artery surgery and lower limb revascularisation under the care of the Vascular Surgery team
2. Willing and able to give informed written consent

Exclusion Criteria:

1. Those unable to give informed written consent
2. Those <18 years of age
3. In the opinion of the investigator unable or unwilling to comply with the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients attending Vascular Surgery department for aortic aneurysm repair, carotid artery surgery and lower limb revascularisation.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between electronic Frailty Index and survival and complication rate. | 6 months
  Survival and rate of complication correlated with the pre-operative frailty score (electronic Frailty Index).
Correlation between Q Mortality Index and survival and complication rate. | 6 months
  Survival and rate of complication correlated with the pre-operative frailty score (Q Mortality Index).
Correlation between ACS Risk Calculator Score and survival and complication rate. | 6 months
  Survival and rate of complication correlated with the pre-operative frailty score (ACS Risk Calculator).
Correlation between V-Possum and survival and complication rate. | 6 months
  Survival and rate of complication correlated with the pre-operative frailty score (V-Possum).

SECONDARY OUTCOMES:
Activity Levels Pre and Post Surgery as measured by the General Practice Physical Activity Questionnaire | 6 months
  General Practice Physical Activity Questionnaire will be used to assess patient reported activity before and after surgery.
Quality of Life Pre and Post Surgery as measure by the EuroQoL EQ-5D questionnaire | 6 months
  EuroQol EQ-5D Quality of Life questionnaire will be used to assess patient reported quality of life before and after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Alun H Davies, DM FRCS, Study Chair — Imperial College London
Locations (2):
- United Kingdom (2):
  - Imperial College London, London
  - Imperial College Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be allowed to be shared on completion.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 3 years for 5 years
Access Criteria: Health researcher for non-commerical research